CLINICAL TRIAL: NCT01997489
Title: Ophthalmic Findings During 10-year Enzyme Substitution of Danish Fabry Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor, chief physician, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fabry-Eyes-13; RH-F-2013 (Other: Rigshospitalet)
Record Dates: First submitted 2013-11-18; First posted 2013-11-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Fabry Disease
Keywords: Eye; Fabry; vessels
MeSH Terms: conditions — Fabry Disease | interventions — Enzyme Replacement Therapy; agalsidase alfa; agalsidase beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fabry patients during treatment (Experimental): 39 patients with Fabry disease having had baseline examinations of the eyes were assessed also at follow-up 10 years after enzyme replacement therapy
  Interventions: Drug: Enzyme replacement

INTERVENTIONS:
Drug: Enzyme replacement — Observational study of current treatment and with no comparative groups
  Other Names: Replagal; Fabrazyme

SUMMARY:
Fabry disease is a recessively inherited disorder due to systemic storage of abnormal metabolites (ceramide trihexocide, in particular) caused by lack of the lysosomal enzyme α-galactosidase. Though X-linked, in patient series there are often equal numbers of males (hemizygotes ) and females (heterozygotes, probably caused by a mutation in one allele and an inactivation on the other allele in the X chromosomes), and many clinical features are shared.

Abnormal storage in endothelial and smooth muscle cells explains morbidity, including a shortened life expectancy. This is due to age dependent ischaemic manifestations that affect heart, kidney and brain. Angiofibroma is an early cutaneous manifestation, and painful acro-paresthesias express juvenile neuropathy.

Cornea verticillata is an almost obligate ophthalmic finding. The brown-yellow Bowman membrane related corneal deposits and teleangiectatic conjunctival vessels are early ophthalmic slit-lamp markers of the disorder; further there can be subtle lens opacities. Fundus vessel tortuosity is observed in many patients, in particular of the retinal venules, but best corrected visual acuity (BCVA) is usually normal.

After the introduction of enzyme substitution therapy in 2001, ophthalmic examinations were scheduled as regular part of the general evaluation of the Fabry patients at Rigshospitalet, Denmark. A 10-year ophthalmic state of arts was part of oral presentations at a Copenhagen conference in December 2011. In contrast to the common occurrence of systemic vascular sequels, only one patient in the series had suffered severe visual loss; this was unilateral and occurred years before institution of the enzyme therapy. In 2013, however, another young male presented a similar retinal event. Sporadic cases of visual loss are reported in the literature, but in larger Fabry series ocular vascular catastrophes appear the exception to the rule.

Following the introduction of enzyme substitution, we found it of interest to present our nationwide Danish experience. We focused on retinal vessel morphology and the relation to systemic morbidity.

DETAILED DESCRIPTION:
Fabry disease is a recessively inherited disorder due to systemic storage of abnormal metabolites (ceramide trihexocide, in particular) caused by lack of the lysosomal enzyme α-galactosidase. Though X-linked, in patient series there are often equal numbers of males (hemizygotes ) and females (heterozygotes, probably caused by a mutation in one allele and an inactivation on the other allele in the X chromosomes), and many clinical features are shared (Cox 2005).

Abnormal storage in endothelial and smooth muscle cells explains morbidity, including a shortened life expectancy (Frost & Tanaka 1966; Desnick et al. 1976; deVeber et al.1992; Hughes & Mehta 2005; Nguyen et al. 2005; Sodi et al. 2007). This is due to age dependent ischaemic manifestations that affect heart, kidney and brain. Angiofibroma is an early cutaneous manifestation, and painful acro-paresthesias express juvenile neuropathy (Cox 2005; Cleary et al. 2005).

Cornea verticillata is an almost obligate ophthalmic finding. The brown-yellow Bowman membrane related corneal deposits and teleangiectatic conjunctival vessels are early ophthalmic slit-lamp markers of the disorder; further there can be subtle lens opacities. Fundus vessel tortuosity is observed in many patients, in particular of the retinal venules, but best corrected visual acuity (BCVA) is usually normal (Ballantyne & Michaelson 1970; Lou et al. 1970; Sher et al. 1979; Utsumi et al. 2009).

After the introduction of enzyme substitution therapy in 2001, ophthalmic examinations were scheduled as regular part of the general evaluation of the Fabry patients at Rigshospitalet, Denmark. A 10-year ophthalmic state of arts was part of oral presentations at a Copenhagen conference in December 2011. In contrast to the common occurrence of systemic vascular sequels, only one patient in the series had suffered severe visual loss; this was unilateral and occurred years before institution of the enzyme therapy (Andersen et al. 1994). In 2013, however, another young male presented a similar retinal event. Sporadic cases of visual loss are reported in the literature (Sher et al. 1978,1979; Tuupurainen et al. 1981; Sakkuraba et al. 1986; Utsumi et al. 2009), but in larger Fabry series ocular vascular catastrophes appear the exception to the rule (Orssaud et al. 2003; Hughes & Mehta 2005; Nguyen et al. 2005; Sodi et al. 2007; Utsumi et al. 2009)).

Following the introduction of enzyme substitution, we found it of interest to present our nationwide Danish experience. We focused on retinal vessel morphology and the relation to systemic morbidity.

ELIGIBILITY:
Inclusion Criteria:

* All Danish patients with Fabry disease before starting therapy

Exclusion Criteria:

* Missing values for eye examination at baseline or follow-up

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2001-09; Primary Completion 2013-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
cornea vercillitata | change from baseline to 10 years
  Eye examination of 39 Fabry patients before starting therapy with enzyme replacement and after 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Ulla Feldt-Rasmussen, Copenhagen, Capital Region
  - National University Hospital, Department of Medical Endocrinology, Copenhagen